CLINICAL TRIAL: NCT01749254
Title: Novel Imaging Approaches To Identify Unstable Coronary Plaques
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/R/CAR/13; ETM/160 (Other Grant/Funding Number: Chief Scientist Office)
Record Dates: First submitted 2012-11-30; First posted 2012-12-13 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease
Keywords: Culprit plaques; Vulnerable Plaques; PET; calcification; inflammation
MeSH Terms: conditions — Coronary Artery Disease; Calcinosis; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute Coronary Syndrome: 40 patients admitted with ACS (NSTEMI/STEMI) will be recruited undergo 18F NaF PET, 18F FDG and CTCA within 1 month of the event.
- Stable angina cohort: 40 patients with previously diagnosed coronary artery disease and listed to undergo elective coronary angiogram will be recruited. VH-IVUS will be attempted in all patients. Selected patients will undergo PET scan after stent implantation.

SUMMARY:
Cardiovascular disease is the leading cause of death in Scotland and the Western World. Approaches to improve the identification of vulnerable or ruptured coronary atherosclerotic plaques are urgently needed to help risk stratification, to identify patients for intensive therapies, and to provide novel biomarkers for the development of anti-atherosclerotic drug interventions. Using positron emission tomography, we have recently shown that sodium 18-fluoride uptake holds major promise as a novel marker of plaque vulnerability and rupture. Here we wish to characterise coronary atherosclerotic plaque using 128-multidetector computed tomography combined with 18-fluorodeoxyglucose and sodium 18-fluoride positron emission tomography and Virtual histology-intravascular ultrasound in 80 patients with stable and unstable coronary artery disease. This has the potential to provide an innovative and highly valuable translational model with which to test novel therapeutic interventions targeted at reducing atheroma and plaque rupture. This could have major implications for the future treatment of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

Age > or = 50 yrs. Patients with Acute coronary syndromes or stable coronary artery disease.

Exclusion Criteria:

Insulin dependent diabetes Inability or unwillingness to undergo computed tomography scanning Severe renal failure (serum creatinine >250 µmol/L or estimated glomerular filtration rate <30 mL/min) Known contrast allergy Inability to give informed consent. Females in child bearing age will undergo pregnancy test if pregnancy suspected.

Participation in other research studies requiring exposure to further radiation (over and above mentioned in this study).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit two populations of 40 patients each. The first population will be patients with known stable coronary heart disease. They will have previously documented and angiographically proven coronary artery disease (≥70% luminal stenosis of a major epicardial vessel). The second population will be patients with a recent (within 30 days) acute myocardial infarction defined by the Universal definition of myocardial infarction. The culprit plaque will be defined according to the invasive coronary angiogram appearances, electrocardiogram and clinical features by two cardiologists blinded to the results of positron emission tomography.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Patients with ACS have focal 18F-NaF uptake and high tissue to background ratio(TBR) and standardised uptake values (SUV) in the culprit vessels. | Within 1 month of index event
  Using PET/CT, the investigators will assess if there is presence of focal uptake at the areas of plaque ruptures in patients presenting with ACS. Standardised uptake values and Tissue to Background ratios of the culprit vessels with be compared with non-culprit lesions.
What are the morphological characteristics of plaque with high 18F-NaF tissue to background ratio or standardised uptake value | 1 month
  Using VH-IVUS, the investigators will look at the morphological characteristics of plaques that have higher SUVs and TBRs. Additional information about the plaque characteristics will be derived from CT coronary angiogram

SECONDARY OUTCOMES:
Is there a co-relation between the two PET/CT tracers(18FDG and 18F NaF) as measured as Tissue to background ratio or standardised uptake value. | 1 month

OTHER OUTCOMES:
Is there a difference between the coronary and aortic TBR/SUVs in stable and unstable patients | 1 month
  The investigators will look for differences in activity in stable angina and ACS patients using 18F-NaF and 18F-FDG
Will patients with higher 18F-NaF uptake as measured by SUV/TBR will have higher levels of cardiac biomarkers such as hsCRP or Troponin | 1 year
  Blood collected from volunteers in the study will be analysed for inflammatory biomarkers such as hsCRP and Troponin

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Imaging Centre/ NHS LOTHIAN, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Result] Joshi NV, Toor I, Shah AS, Carruthers K, Vesey AT, Alam SR, Sills A, Hoo TY, Melville AJ, Langlands SP, Jenkins WS, Uren NG, Mills NL, Fletcher AM, van Beek EJ, Rudd JH, Fox KA, Dweck MR, Newby DE. Systemic Atherosclerotic Inflammation Following Acute Myocardial Infarction: Myocardial Infarction Begets Myocardial Infarction. J Am Heart Assoc. 2015 Aug 27;4(9):e001956. doi: 10.1161/JAHA.115.001956. PMID 26316523